CLINICAL TRIAL: NCT07036042
Title: Clinical Characteristics of Patients With Anti-Collapsin Response Mediator Protein 2 Antibodies in Encephalitis or Encephalomyelitis
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-180
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autoimmune encephalitis (AE) is an important autoimmune neurological disease, and its clinical manifestations, treatment and prognosis are closely related to the type of pathogenic antibodies. However, due to the limited antibody spectrum and the unclear pathogenic mechanism, the disease is difficult to diagnose and treat, and the morbidity and mortality rates are high. In a previous study, we found that anti-CRMP2 antibodies were AE-specific autoantibodies, adding a new member to the AE antibody spectrum and thus defining a new class of AEs, anti-CRMP2 encephalitis. However, due to the limited number of cases, its clinical characteristics such as incidence, concomitant diseases, imaging manifestations, treatment effects and prognosis are not yet clear. This study plans to conduct large-scale anti-CRMP2 antibody screening in critically ill patients with suspected neurological autoimmune diseases in our hospital, and compare the clinical differences between anti-CRMP2 encephalitis and other known AEs and non-autoimmune encephalitis.

ELIGIBILITY:
The inclusion criteria for patients are illustrated: 1) patients admitted to the Department of Neurology,or the Neurocritical Unit (NCU) of Nanfang Hospital, Southern Medical University, between January 2017 and November 2019; 2) patients with suspected immune-mediated encephalopathy (altered consciousness persisting for more than 24 hours) or myelopathy. This included cases of encephalopathy suspected to be autoimmune, infectious or metabolic as well as encephalopathy with unclear etiology; 3) patients with remaining serum and/or cerebrospinal fluid (CSF) samples available for immunoreaction analysis using tissue-based assay (TBA) and cell-based assay (CBA). All samples were the first obtained from patients after hospitalization, prior to initiating treatment at our hospital. Some patients, however, may have received treatment at other hospitals before being transferred here.

The exclusion criteria were: 1) loss to follow-up; 2) incomplete data; 3) encephalopathy resulting from toxic, traumatic, anoxic/hypoxic, genetic, or endocrine causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Neurology, Nanfang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Antibodies CRMP2 detected in blood or cerebrospinal fluid | 2024.12

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All participants' data are confidential.